CLINICAL TRIAL: NCT03459521
Title: Efficacy of Hepatitis B Virus Vaccines HBVaxpro40© and Fendrix© in Patients With Chronic Liver Disease in Clinical Practice.
Brief Title: Efficacy of HBVaxpro40© and Fendrix© in Patients With Chronic Liver Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Diana Horta-Sangenis, Principal Investigator, Corporacion Parc Tauli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HMT2
Record Dates: First submitted 2017-06-19; First posted 2018-03-09 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Liver Disease Chronic; Hepatitis B Virus
MeSH Terms: conditions — Hepatitis B | interventions — Fendrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fendrix HBV vaccine or HBVaxpro 40 (Experimental): Drug: Fendrix Fendrix suspension for injection GlaxoSmithKline Route of administration, dose regimen: Intra-muscular Dose: 20mcg of Hepatitis B Surface Antigen per vaccination at baseline, 1, 2 and 6 months.
  Drug: HBVaxpro 40 Sanofi Pasteur MSD Route of administration, dose regimen: Intra-muscular Dose: 40mcg of Hepatitis B Surface Antigen per vaccination at baseline, 1 and 6 months.
  Interventions: Biological: Fendrix or HBVAXPRO 40

INTERVENTIONS:
Biological: Fendrix or HBVAXPRO 40 — To administer hepatitis B virus vaccines in patients with chronic liver disease that have not been previously vaccinated.

SUMMARY:
Background: Cirrhotic patients have an increased risk of infections. In these patients is important to prevent hepatitis B virus (HBV) infection, as it may cause a deterioration of liver function. However, HBV vaccine efficacy in this group of patients is lower than in healthy population. Despite increasing standard doses to double doses or administering an accelerated pattern, the response to HBV vaccination remains suboptimal. For this reason, an alternative strategy may be using vaccines with novel adjuvants such as Fendrix® or the recombinant vaccine HBVAXPRO®.

Aim: To assess the adjuvanted HBV vaccine (Fendrix ®) efficacy in patients with chronic liver disease and to understand the kinetics of anti-HBs titers over time in patients who respond to vaccination.

Methods: Prospective and multicenter study. Serological markers of HBV will be assessed prospectively in consecutive patients with non-cirrhotic liver disease (permanent abnormal liver blood tests > six months; elastogram ≥8 kilopascal (kPa); serum markers of fibrosis (APRI or FIB-4 ≥ F2); ultrasound changes suggesting chronic liver disease) and cirrhotic patients (diagnosed by liver biopsy and/or non-invasive methods: clinical, blood tests and ultrasound). Seronegative patients will receive four doses of Fendrix ® at 0,1, 2 and 6 months. Antibodies against HBV superficial antigen (anti-HBs) will be determined at 2 months +/- 10 days, six months and one year after having received the fourth dose of the vaccine (to see kinetics). The study will differentiate between responders and non-responders to the vaccine: adequate immunity to HBV will be defined as anti-HBs higher than > 10mUI/mL (standard definition of seroconversion) and> 100mUI/mL. Investigators will evaluate the factors that influence the response, kinetics and safety of the vaccination in patients with chronic liver disease and cirrhosis.

DETAILED DESCRIPTION:
Intervention: Serological markers of HBV will be assessed prospectively in consecutive non-cirrhotic liver disease or cirrhotic patients. Seronegative patients willing to participate will sign a written informed consent and will receive four doses of 20 µg Fendrix ® at 0,1, 2 and 6 months or HBVAXPRO® at 0,1 and 6 months, depending on availability. Antibodies against HBV superficial antigen (anti-HBs) will be determined at 2 months +/- 10 days, six and twelve months after having received the fourth dose of the vaccine (to see kinetics). The study will differentiate between responders and nonresponders to the vaccine: adequate immunity to HBV will be defined as anti-HBs higher than > 10mUI/mL (standard definition of seroconversion) and > 100mUI/mL. Adverse events will be assessed throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Chronic liver disease patients -non-cirrhotic and cirrhotic- diagnosed by liver biopsy and / or non-invasive methods (by standard clinical, analytical and ultrasound crite-ria)
* Negative hepatitis B surface antigen (HBs Ag) and antibody to hepatitis B core antigen (anti-HBc).

Exclusion Criteria:

* Allergy to vaccine components (sodium chloride, aluminium phosphate)
* Active or past HBV infection
* Patients previously vaccinated against HBV (regardless of response)
* Child-Pugh C
* Conditions that cause immunosuppression (HIV infection, chronic renal failure, active neoplasia)
* Pregnancy or breastfeeding
* Non-immunized HAV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
The proportion of individuals seroconverting with Hepatitis B surface antibody titres of > 10 and > 100 UI/ml. | 8 months

SECONDARY OUTCOMES:
Number of Participants With Vaccine-Related Adverse Events as Assessed by CTCAE v4.0 | 8 months

OTHER OUTCOMES:
The durability of anti-HBs titers over time in patients who respond to vaccination. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Diana Horta, Principal Investigator — Corporacion Parc Tauli
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona/Spain, Spain

IPD SHARING:
Plan to Share IPD: No